CLINICAL TRIAL: NCT04702880
Title: A Randomized, Open-label Phase 2 Clinical Trial of BMS-986012 in Combination With Carboplatin, Etoposide, and Nivolumab as First-line Therapy in Extensive-stage Small Cell Lung Cancer
Brief Title: A Study of BMS-986012 in Combination With Carboplatin, Etoposide, and Nivolumab as First-line Therapy in Extensive-stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA001-050; 2020-001863-10 (EudraCT Number); U1111-1250-4427 (Registry Identifier: WHO)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: BMS-986012; Carboplatin; Etoposide; Extensive-stage small cell lung cancer; Fucosyl; Nivolumab; Targeted SCLC therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Carboplatin + Etoposide + Nivolumab + BMS-986012 (Experimental)
  Interventions: Biological: BMS-986012; Drug: Carboplatin; Drug: Etoposide; Biological: Nivolumab
- Arm B: Carboplatin + Etoposide + Nivolumab (Experimental)
  Interventions: Drug: Carboplatin; Drug: Etoposide; Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986012 — Specified dose on specified days
  Other Names: Fucosyl-GM1 Antibody
  Arms: Arm A: Carboplatin + Etoposide + Nivolumab + BMS-986012
Drug: Carboplatin — Specified dose on specified days
Drug: Etoposide — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to demonstrate that treatment with BMS-986012 in combination with carboplatin, etoposide, and nivolumab will have acceptable safety and tolerability and will improve progression-free survival compared with carboplatin, etoposide, and nivolumab alone in newly diagnosed participants with extensive-stage small cell lung cancer (ES-SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented extensive-stage small cell lung cancer (ES-SCLC) and extensive-stage disease (American Joint Committee on Cancer, 8th edition, Stage IV [T any, N any, M1a, M1b, or M1c], or T3-4 due to multiple lung nodules that are too extensive or tumor or nodal volume that is too large to be encompassed in a tolerable radiation plan)
* Participants taking part in the separate PET tracer sub-study must provide a fresh tumor biopsy from any disease site (primary or metastatic)
* Archived tumor specimens, in the form of blocks or sectioned slides, are mandatory for all participants except those participating in the separate PET tracer sub-study for whom the archived tumor specimen is optional
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1
* At least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria
* Adequate hematologic and end organ function
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are pregnant or breastfeeding. Japan only: participation in the study is not allowed even if breastfeeding is suspended
* Prior chemotherapy, radiation therapy, or biologic therapy for SCLC. Previously treated limited stage SCLC (LS-SCLC) participants are also excluded
* Symptomatic brain or other central nervous system (CNS) metastases
* Paraneoplastic autoimmune syndrome requiring systemic treatment
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, idiopathic pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan
* Grade ≥ 2 peripheral sensory neuropathy at study entry
* Significant uncontrolled cardiovascular disease
* Active, known or suspected autoimmune disease or inflammatory disorder

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years and 100 days
Incidence of serious adverse events (SAEs) | Up to 2 years and 128 days
Incidence of AEs leading to discontinuation | Up to 2 years and 128 days
Incidence of deaths | Up to 2 years and 128 days
Progression-free survival (PFS) by blinded independent central review (BICR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | Up to 2 years

SECONDARY OUTCOMES:
Progression-free survival rate (PFSR) | 6 and 12 months
  PFS by BICR based on RECIST v1.1 criteria
PFS by investigator based on RECIST v1.1 criteria | Up to 2 years
PFSR | 6 and 12 months
  PFS by investigator based on RECIST v1.1 criteria
Objective response rate (ORR) based on RECIST v1.1 criteria | Up to 2 years
Time to response (TTR) based on RECIST v1.1 criteria | Up to 2 years
Duration of response (DOR) based on RECIST v1.1 criteria | Up to 2 years
Overall survival (OS) | Up to 3 years
  By arm
Overall survival rate (OSR) | Up to 3 years
  By arm
Immunogenicity of BMS-986012 measured by assessment of the presence of specific anti-drug antibodies (ADAs) to BMS-986012 (i.e. incidence of positive ADAs) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (8):
  - Local Institution - 0075, Birmingham, Alabama
  - Local Institution - 0022, Hackensack, New Jersey
  - Local Institution - 0002, Durham, North Carolina
  - Local Institution - 0060, Cincinnati, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution - 0067, Cleveland, Ohio
  - Local Institution - 0081, Nashville, Tennessee
  - Local Institution, Dallas, Texas
- Australia (4):
  - Local Institution - 0003, Westmead, New South Wales
  - Local Institution - 0023, Greenslopes, Queensland
  - Local Institution - 0001, Malvern, Victoria
  - Local Institution - 0004, Murdoch, Western Australia
- Belgium (3):
  - Local Institution - 0051, Charleroi, Hainaut
  - Local Institution - 0034, Ghent
  - Local Institution - 0050, Liège
- Canada (2):
  - Local Institution - 0012, Edmonton, Alberta
  - Local Institution - 0064, Brampton, Ontario
- Greece (3):
  - Local Institution - 0045, Heraklion, Irakleío
  - Local Institution - 0036, Athens
  - Local Institution - 0038, Athens
- Italy (3):
  - Local Institution - 0030, Peschiera del Garda
  - Local Institution - 0031, Pisa
  - Local Institution - 0029, Rozzano
- Japan (4):
  - Local Institution - 0073, Sendai, Miyagi
  - Local Institution - 0070, Ōsaka-sayama, Osaka
  - Local Institution - 0069, Takatsuki, Osaka
  - Local Institution - 0077, Ina-machi, Saitama
- Netherlands (3):
  - Local Institution - 0039, Amsterdam, North Holland
  - Local Institution - 0066, Arnhem
  - Local Institution - 0040, Groningen
- Poland (2):
  - Local Institution - 0049, Gdansk
  - Local Institution - 0048, Lodz
- Romania (3):
  - Local Institution - 0043, Bucharest
  - Local Institution - 0042, Cluj-Napoca
  - Local Institution - 0041, Craiova
- Spain (4):
  - Local Institution - 0007, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0021, Madrid
  - Local Institution - 0005, Majadahonda
  - Local Institution - 0006, Málaga

REFERENCES:
- [Derived] Chu Q, Leighl NB, Surmont V, van Herpen C, Sibille A, Markman B, Clarke S, Juergens RA, Rivera MA, Andelkovic V, Rudin CM, Snow S, Kim DW, Sanatani M, Lin H, Sanghavi K, Tannenbaum-Dvir S, Basciano P, Lathers D, Urbanska K, Kollia G, He C, DiPiero A, Liu Y, Ready N. BMS-986012, an Anti-Fucosyl-GM1 Monoclonal Antibody as Monotherapy or in Combination With Nivolumab in Relapsed/Refractory SCLC: Results From a First-in-Human Phase 1/2 Study. JTO Clin Res Rep. 2022 Aug 27;3(11):100400. doi: 10.1016/j.jtocrr.2022.100400. eCollection 2022 Nov. PMID 36275912
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04702880.html